CLINICAL TRIAL: NCT07056036
Title: Safety and Efficacy of BTL-699-2 for the Improvement in Willpower, Self-control & Food Cravings
Brief Title: EXOMIND (BTL-699-2) for the Improvement in Willpower & Food Cravings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTL-699_CTUS200
Record Dates: First submitted 2025-06-10; First posted 2025-07-09 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-06

CONDITIONS: Self-Control; Food Cravings
Keywords: self-control; willpower; food cravings; rTMS; ExoTMS; EXOMIND
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active treatment with BTL-699-2 (Experimental): Participants will receive BTL-699-2 treatments with an intensity of up to 70% of their motor threshold.
  Interventions: Device: ActiveTreatment with BTL-699-2
- Sham treatment with BTL-699-2 (Sham Comparator): Participants will receive BTL-699-2 treatments with an intensity of 5% of their motor threshold.
  Interventions: Device: Sham Treatment with BTL-699-2

INTERVENTIONS:
Device: ActiveTreatment with BTL-699-2 — Participants will receive six transcranial magnetic stimulation treatments with the BTL-699-2 device over the left dorsolateral prefrontal cortex. The intensity will be adjusted according to the subject's feedback, up to 70% of the individual's motor threshold. The treatments will be spaced 3 - 7 days apart.
  Other Names: EXOMIND (BTL-699-2) ActiveTreatment
  Arms: Active treatment with BTL-699-2
Device: Sham Treatment with BTL-699-2 — Participants will receive six transcranial magnetic stimulation treatments with the BTL-699-2 device over the left dorsolateral prefrontal cortex. The intensity will se to 5% of the individual's motor threshold. The treatments will be spaced 3 - 7 days apart.
  Other Names: EXOMIND (BTL-699-2) ShamTreatment
  Arms: Sham treatment with BTL-699-2

SUMMARY:
The goal of this clinical trial is to evaluate if the treatment with ExoMIND (BTL-699-2) device is able to improve willpower, self-control and food cravings in adults above the age of 22 years. The main question it aims to answer is:

Does the treatment with EXOMIND (BTL-699-2) device improve willpower, self-control and food cravings?

Participants will be asked to:

* Undergo six treatments
* Complete the Brief Self-control Scale
* Complete the Food Cravings Questionnaire - Trait
* Complete the Therapy Comfort Questionnaire
* Complete the Subject Satisfaction Questionnaire

DETAILED DESCRIPTION:
This study uses a prospective, multi-center, two-arm, sham-controlled, single-blinded interventional study design.

The subjects will be enrolled and assigned to two experimental study arms: the active group (Group A) and the sham group (Group B), in a ratio of 3:1. All enrolled participants will be treated (either active or sham) with the BTL-699-2 device. Group A will receive rTMS treatment with an intensity of up to 70% of their MT, while Group B will receive rTMS treatment with an intensity of 5% of their MT. Six (6) treatments will be delivered, 3-7 days apart. Examination for possible adverse effects will be conducted after each treatment.

The Brief Self-Control Scale and the Food Cravings Questionnaire - Trait (FCQ-T) will be administered to the subjects before the first treatment, after the last treatment, and at the two follow-up visits-1 month and 3 months after the final session.

The Therapy Comfort Questionnaire will be administered after the last treatment, while the Subject Satisfaction Questionnaire will be given after the last treatment and at both follow-up visits.

The total expected duration of subject participation, from the baseline visit to study completion, is approximately five months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 22 years
* Ability to determine the motor threshold of the participant. The participant's motor threshold could be established as the minimum stimulus required to induce contraction of the right thumb
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure for the improvement of willpower and self-control and rI eduction of food cravings, including non-invasive brain stimulation treatments other than the study procedure during study participation
* Subjects willing and able to maintain their regular (pre-procedure) exercise regimen without affecting significant change in either direction during study participation
* Willingness to comply with study instructions and to return to the clinic for the required visits
* Women of child-bearing potential* are required to use birth control measures during the whole duration of the study
* If applicable, subjects will be maintained on pre-study prescribed medications at a stable therapeutic dosage for at least 2 months prior to study entry

Exclusion Criteria:

* Electronic implants (Implanted stimulator devices in or near the head - rTMS devices are contraindicated for use in patients who have active or inactive implants (including device leads), deep brain stimulators, cochlear implants, ocular implant, and vagus nerve stimulators, implanted devices such as cardiac pacemakers, defibrillators, neurostimulators. Contraindicated use could result in serious injury or death.
* Metallic, conductive, ferromagnetic or other magnetic sensitive implants/objects in the head or within 30 cm of the treatment coil (examples include implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, jewelry and hair barrettes) with some exceptions in the mouth as standard amalgam dental fillings, single post dental implants, and dental bridge work. Failure to follow this restriction could result in serious injury or death.
* Drug pump(s)
* Application in the heart area
* Persons with a tendency to seizure (hypotonic, epileptic), or a personal history of epilepsy
* Ongoing anticoagulation therapy
* Ongoing severe or life-threatening condition
* Pulmonary insufficiency
* Heart disorders
* Renal insufficiency
* Decompensated* hemorrhagic conditions, blood coagulation disorders, cardiovascular diseases
* Malignant or benign tumor
* Fever
* Ongoing pregnancy or nursing
* Ongoing intake disorders such as bulimia or anorexia
* Diagnosis of major depression, depression, post-traumatic stress disorder, psychotic disorder or current psychotic symptoms, bipolar disorder, obsessive-compulsive disorder, borderline personality disorder
* Personal history of syncope (except the reflex syncope)
* Vascular, traumatic, tumoral, infectious, or metabolic lesion of the brain, even without a history of seizure, and without anticonvulsant medication
* Withdrawal from one of the following drugs could form a relative hazard for the application of rTMS due to the resulting significant seizure threshold lowering potential: (e.g. alcohol, barbiturates, benzodiazepines, meprobamate, chloralhydrate etc.)
* Systemic infection
* Patients with a broad range of neuropsychiatric diseases are at elevated risk for seizures. Essentially all neurologic conditions with structural cerebral damage (e.g. stroke, multiple sclerosis, traumatic brain injury, Alzheimer's and other neurodegenerative diseases, meningoencephalitis or intracerebral abscess, parenchymal or leptomeningeal cancers)
* History of hyponatremia, hypocalcemia, hypomagnesemia, hypoglycemia, hyperglycemia, renal failure/uremia, liver failure
* History of tendency for raised blood concentrations of pro-convulsant medications due to reduced clearance
* Immunosuppressive therapy with cyclosporine, tacrolimus and other agents that can cause the posterior reversible leukoencephalopathy syndrome
* The use of methamphetamine, barbiturates, cocaine metabolites, opiates and phencyclidine 72 hours before the therapy
* Contradictions for the testing used in the trial, for example, the motor threshold cannot be found or quantified.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Assessment of Change in Willpower and Self-control | 15 months
  The change in the score obtained from the Brief Self-Control scale will be recorded. The questionnaire will be administered at the baseline visit, after the last treatment, at the 1-month and 3-month follow-up visits. The score ranges from 13 to 65 and higher scores indicate a higher level of self-control. An improvement is defined as an increase in score.

SECONDARY OUTCOMES:
Assessment of Change in Food Cravings | 15 months
  The change in the score obtained from the Food Cravings Questionnaire - Trait (FCQ-T) will be recorded. The questionnaire will be administered at the baseline visit, after the last treatment, at the 1-month and 3-month follow-up visits. The score ranges from 39 to 234 and higher scores indicate more frequent and intense experiences of food craving in general. An improvement is defined as a decrease in score.
Assessment of Satisfaction | 15 months
  Subject Satisfaction with treatment outcomes will be assessed using 5-point Likert Scale Subjects Satisfaction Questionnaire. The questionnaire will be administered after the last treatment, at the 1-month and 3-month follow-up visits. Responses to questions about satisfaction with the treatment outcomes will range from "strongly disagree" (1 point) to "strongly agree" (5 points). A higher score for each statement indicate better outcomes.
Assessment of Therapy Comfort | 15 months
  Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. The Therapy Comfort questionnaire will be administered after the last treatment. Therapy Comfort questionnaire consists of the question "I found the treatment comfortable", to which responses are based on a 5-point Likert scale (1 = "strongly disagree", and 5 = "strongly agree"). A higher score for the statement "I found the treatment comfortable" indicate higher therapy comfort.
Assessment of Pain During Therapy | 15 months
  The Therapy Comfort Questionnaire will be used to evaluate pain experienced during treatment sessions. It will be administered after the final treatment. The questionnaire includes a 10-point Numeric Analog Scale for pain (0 = no pain, 10 = worst possible pain). Lower scores on the Numeric Analog Scale indicate lower levels of pain.
Incidence of Treatment-related Adverse Events | 15 months
  Monitoring of adverse reactions and side effects will be performed for the evaluation of safety of the treatment with the BTL-699-2 device for the improvement of well-being and to identify side effects and adverse events associated with the study treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Aria Integrative Health, Denver, Colorado
  - A New You Wellness, Miami, Florida
  - Cady Wellness Institute, Newburgh, Indiana
  - Jiva Med Spa, Columbus, Ohio